CLINICAL TRIAL: NCT01501266
Title: Faslodex Specific Clinical Experience Investigation for Long-term Use
Brief Title: Faslodex Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6997C00008
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: postmenopausal breast cancer; Faslodex; cohort
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Faslodex

SUMMARY:
The purpose of this study is to confirm the safety profile such as the frequency of serious adverse events or any unexpected adverse events and overall efficacy of Faslodex for long term treatment in daily clinical practice.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Faslodex for the first time due to postmenopausal breast cancer

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Faslodex for the first time due to postmenopausal breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions. | 1 year
Incidence of serious adverse events. | 1 Year

SECONDARY OUTCOMES:
Incidence of adverse drug reactions with injection site reaction, thromboembolic events and hepatic impairment | 1 year
Progression-free survival | 6 month
Progression-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, Study Director — AstraZeneca KK
Locations (43):
- Japan (43):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: CSR_Synopsis_D6997C00008 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=590&filename=CSR_Synopsis_D6997C00008.pdf
- See also: D6997C00008Fulvestrant_Specific_Clinical_Experience_Investigation_Protocol_redacted_23February2016 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=590&filename=D6997C00008Fulvestrant_Specific_Clinical_Experience_Investigation_Protocol_redacted_23February2016.pdf